CLINICAL TRIAL: NCT03323918
Title: Parent-implemented Intervention for Children With ASD: Effect on Social Communication and Brain Activation
Brief Title: ImPACT Intervention for Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRAINVIEW/ESR14
Record Dates: First submitted 2017-10-02; First posted 2017-10-27 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Group 1 will receive the intervention specifically targeting social-communicative abilities (Project ImPACT).
  Group 2 will receive a generic intervention, that will not focus on social-communicative skills.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators who are involved in the testing sessions and data analysis are blind to group assignment. An investigator which is not directly involved in participant testing or data analysis takes care of the randomisation, and coordinates it with the home guidance centers that administer the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImPACT (Experimental): Project ImPACT will be provided in 18 weekly intervention sessions, during which parents will learn how to stimulate their children's social imitation, social engagement, language and play skills. First, parents are taught techniques that promote interaction with the child (one technique per session, through demonstration and coaching). In the second half of the intervention, parents are taught direct teaching techniques, e.g., to promote language or play, again by means of demonstration and coaching. After completion of the program, families will receive guidance every 2-3 weeks for an additional 12 weeks, during which the support will generally not focus on social-communicative abilities, although ImPACT follow-up sessions might be given if necessary.
  Interventions: Other: ImPACT
- TAU (Active Comparator): Treatment as usual (TAU) will be provided at the typical frequency, which is every 2-3 weeks. TAU can include targeting eating and sleeping problems, adaptive skills, or other goals. TAU will not include forms of intervention explicitly targeting social communicative skills. However, limited guidance on social communication development can be given if explicitly asked by parents.
  Interventions: Other: TAU

INTERVENTIONS:
Other: ImPACT — Teaching parents to train social communicative skills as outlined in arm description.
  Arms: ImPACT
Other: TAU — TAU can include targeting eating and sleeping problems, adaptive skills, or other goals.
  Other Names: Treatment as usual
  Arms: TAU

SUMMARY:
This randomised-controlled trial will assess the effect of an early intervention on the social-communicative abilities and brain activity of preschoolers with autism spectrum disorder (ASD). The children´s social-communicative abilities and the related brain activity will be evaluated at three time points: before the start of the intervention (pre-intervention), immediately after its conclusion (post-intervention) and several weeks after its conclusion (follow-up).

DETAILED DESCRIPTION:
Previous research has shown that parent-implemented interventions are effective in improving the social skills of children with autism spectrum disorder (ASD). The aim of the present project is to investigate the brain activity changes that are at the basis of the changes observed in the children's behaviour. More specifically, the investigators will assess the effect of Project ImPACT, a parent-implemented intervention, which teaches parents techniques to stimulate the social-communicative abilities of their children.

The intervention is suitable for preschoolers with a diagnosis of ASD and consists of 18 sessions of maximum 2 hours each, one session per week, delivered by trained therapists of the home guidance services in Flanders. Children with a diagnosis of ASD (or children who are suspected of ASD) between 1,5 and 4 years old and their parents will participate in the study. They will be randomly assigned to the ImPACT intervention or treatment as usual. The investigators will assess the effect of the intervention on the children's social-communicative abilities, and on the neural and biological correlates of these abilities.

The families will be invited to come to the Faculty of Psychology and Pedagogical Sciences at three time points: before the start of the intervention, immediately after the end of the intervention (which is expected to last 18 weeks) and 12 weeks after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* A clinical or working diagnosis of ASD

Exclusion Criteria:

-

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the score of the Early Social Communication Scales (ESCS) | outcome at 18 weeks from start of intervention (post-test)
  Structured observation of interaction with experimenter assessing joint attention. The measure includes continuous measurement of initiation of joint attention (IJA) and behavioural requests (IBR). The measurement of response to joint attention (RJA) is constrained by the numbered of joint attention bids offered by the administer, which is 14 in total. The IJA, IBR, and RJA subsections are considered separately, and the three scores are not combined. An increase in the IJA and RJA scores is interpreted as an improvement. A decrease in IBR, if combined with an increase of IJA, is generally also interpreted as a qualitative improvement of a child's social initiatives.
Change from baseline in the score of a semi-structured social imitation task | outcome at 18 weeks from start of intervention (post-test)
  Unpublished task developed by B. Ingersoll, author of the ImPACT intervention programme. Semi-structured observation of interaction with experimenter. Only the object scale is in use. The score ranges from 0 to 20, with higher scores corresponding to higher social imitation rates.
  Score increase is a positive outcome.
Change from baseline in the score of the Brief Observation of Social Communication Change (BOSCC) | outcome at 18 weeks from start of intervention (post-test)
  Semi-structured observation of interaction with parent and experimenter to assess social communication.
  The test contains 9 items that are meant to capture the quality of a child's social interaction, for which the total scores ranges from 0 to 45, and 3 items describing restricted a repetitive behaviour, which is also part of the ASD symptomatology, the total score of which ranges from 0 to 15. Three additional items are coded to add information on symptoms that might be present although they are not specifically part of the ASD syndrome, and refer to activity level, disruptive behaviour, and anxious behaviours.
  The BOSCC total score consists in the sum of the total score obtained in the first twelve items (ASD specific symptoms), and ranges from 0 to 60, with the three extra items added separately to integrate information.
  In the total and subscale scores, higher scores correspond to more severe symptoms. A decrease in the total score is thus considered a positive outcome.
Change from baseline in electrophysiological event-related potentials in response to voice and non-voice sounds (N1, N2 and P3 effects), measured with EEG | outcome at 18 weeks from start of intervention (post-test)
  EEG activity will be recorded while children watch silent movies and passively listen to voice and non-voice sounds (passive oddball paradigm).
Change from baseline in haemodynamic response function (oxyhaemoglobin and deoxyhaemoglobin concentration in the cerebral cortex) evoked by social attention cues, measured with NIRS (near infrared spectroscopy) | outcome at 18 weeks from start of intervention (post-test)
  Oxy- and deoxyhaemoglobin concentration measured during a task in which an experimenter establishes social and non-social attention conditions while children watch fragments of age-appropriate cartoons.
Change from post-test in the score of the Early Social Communication Scales (ESCS) | follow-up at 12 weeks from end of intervention
  Structured observation of interaction with experimenter assessing joint attention. The measure includes continuous measurement of initiation of joint attention (IJA) and behavioural requests (IBR). The measurement of response to joint attention (RJA) is constrained by the numbered of joint attention bids offered by the administer, which is 14 in total. The IJA, IBR, and RJA subsections are considered separately, and the three scores are not combined.
  Stability (after increase at outcome) or increase in the IJA and RJA scores is interpreted as an improvement. A decrease in IBR, if combined with an increase of IJA, is generally also interpreted as a qualitative improvement of a child's social initiatives.
Change from post-test in the score of a semi-structured social imitation task | follow-up at 12 weeks from end of intervention
  Unpublished task developed by B. Ingersoll, author of the ImPACT intervention programme. Semi-structured observation of interaction with experimenter. Only the object scale is in use. The score ranges from 0 to 20, with higher scores corresponding to higher social imitation rates.
  Score stability (after increase at outcome) or increase is a positive outcome.
Change from post-test in the score of the Brief Observation of Social Communication Change (BOSCC). | follow-up at 12 weeks from end of intervention
  Semi-structured observation of interaction with parent and experimenter to assess social communication. The test contains 9 items that are meant to capture the quality of a child's social interaction, for which the total scores ranges from 0 to 45, and 3 items describing restricted a repetitive behaviour, which is also part of the ASD symptomatology, the total score of which ranges from 0 to 15. Three additional items are coded to add information on symptoms that might be present although they are not specifically part of the ASD syndrome, and refer to activity level, disruptive behaviour, and anxious behaviours. The BOSCC total score consists in the sum of the total score obtained in the first twelve items (ASD specific symptoms), and ranges from 0 to 60, with the three extra items added separately to integrate information. In the total and subscale scores, higher scores correspond to more severe symptoms. Score stability (after decrease at outcome) or decrease is a positive outcome.
Change from post-test in electrophysiological event-related potentials in response to voice and non-voice sounds (N1, N2 and P3 effects), measured with EEG | follow-up at 12 weeks from end of intervention
  EEG activity recorded while children watch silent movies and passively listen to voice and non-voice sounds (passive oddball paradigm).
Change from post-test in haemodynamic response function (oxyhaemoglobin and deoxyhaemoglobin concentration in the cerebral cortex) evoked by social attention cues, measured with NIRS (near infrared spectroscopy) | follow-up at 12 weeks from end of intervention
  Oxy- and deoxyhaemoglobin concentration measured during a task in which an experimenter establishes social and non-social attention conditions while children watch fragments of age-appropriate cartoons.

SECONDARY OUTCOMES:
Change from baseline in the score of the Autism Diagnostic Observational Scale - 2 (ADOS-2) | follow-up at 30 weeks from beginning of intervention
  A standard measure internationally used to identify symptoms of autism. The total score ranges from 0 to 30, with a higher score corresponding to higher symptom severity. The total score results from the sum of two subscales: the Social Affect subscale (SA), with scores ranging from 0 to 22, and the Restricted and Repetitive Behavior one (RRB), with scores ranging from 0 to 8. The ADOS-2 total score is converted through an age-dependednt algorithm to a diagnostic ordinal scale ranging from 0 to 10 (with higher scores indicating higher symptom severity), based on which a diagnostic classification can be formulated (no ASD, ASD, autism).
  A reduction in the total score, as well as in a subscale score, is considered a positive outcome, particularly if this leads to a decrease in the conversion score and/or to a milder diagnostic classification.
Change from baseline in the score of the Mullen Scales of Early Learning (M-SEL) | follow-up at 30 weeks from beginning of intervention
  An age-appropriate measure of cognitive development. It measures a child's IQ on a continuous scale from 49 to 130 points, with the average being 100 points. If the child's IQ is lower than 49 or higher than 130, a general indication of <49 or >130 is given. It also provides an indication of a child's mental age between 0 and 68 months. A growth in mental age over time is considered a neutral outcome. A high growth rate (= the change in months is higher than the number of months actually passed between baseline and follow-up) in a domain where a child initially showed a delay is considered a positive outcome.
Change from baseline in the score of the Vineland screener questionnaire (0-6 years). | outcome at 18 weeks from start of intervention (post-test)
  Questionnaire to assess adaptive skills. The composite score is computed as the sum of subscale scores: communicative skills (0-38), social skills (0-38), everyday skills (0-16), motor skills (0-36). Raw scores can be converted to adaptive age.
  Score increase is a positive outcome.
Change from baseline in the score of the Dutch adaptation of the MacArthur Communicative Development Inventories (NCDI - short form) | outcome at 18 weeks from start of intervention (post-test)
  Parent report of language development (questionnaire). The questionnaire consists of two subsection: a) number of comprehended words (out of 112), b) number of actively used words (out of 112). The two subscales are kept separate, and no composite score is computed.
  The section in use is the 2A section, which is meant for children between 16 and 30 months. Because a number of children in the study are older than 30 months, only the raw scores are taken into account.
  Score increase is considered a positive outcome.
Change from baseline in the score of the Nijmeegse Ouderlijke Stress Index | outcome at 18 weeks from start of intervention (post-test)
  Questionnaire over Parenting stress index developed in Nijmegen. Scores range from 0 to 738, distributed over two main subscales: parent-related stress, maximum score 390, and child-related stress, maximum score 348. Each subscale is composed of subdomains. The parent-related stress is described by competence (0-78), role restriction (0-42), attachment (0-42), depression (0-72), health (0-36), social isolation (0-36), marital relationship (0-42). The child-related stress is described by adaptation (scores: 0-78), temperament (0-60), distractability (0-72), demandingness (0-60), positive reinforcement (0-48), acceptance (0-72). An algorithm converts the subscores and the total score to a descriptive classification of parental stress level (very low, low, below average, average, above average, high, very high). Special norms hold for clinical samples.
  Higher values correspond to higher parental stress. A score reduction is a positive outcome.
Change from post-test in the score of the Vineland screener questionnaire (0-6 years). | follow-up at 12 weeks from end of intervention
  Questionnaire to assess adaptive skills. The composite score is computed as the sum of subscale scores: communicative skills (0-38), social skills (0-38), everyday skills (0-16), motor skills (0-36). Raw scores can be converted to adaptive age.
  Score stability (after increase) or increase is a positive outcome.
Change from post-test in the score of the Dutch adaptation of the MacArthur Communicative Development Inventories (NCDI - short form) | follow-up at 12 weeks from end of intervention
  Parent report of language development (questionnaire). The questionnaire consists of two subsection: a) number of comprehended words (out of 112), b) number of actively used words (out of 112). The two subscales are kept separate, and no composite score is computed.
  The section in use is the 2A section, which is meant for children between 16 and 30 months. Because a number of children in the study are older than 30 months, only the raw scores are taken into account.
  Score stability (after increase at outcome) or increase is considered a positive outcome.
Change from post-test in the score of the Nijmeegse Ouderlijke Stress Index | follow-up at 12 weeks from end of intervention
  Questionnaire over Parenting stress index developed in Nijmegen. Scores range from 0 to 738, distributed over two main subscales: parent-related stress, maximum score 390, and child-related stress, maximum score 348. Each subscale is composed of subdomains. The parent-related stress is described by competence (0-78), role restriction (0-42), attachment (0-42), depression (0-72), health (0-36), social isolation (0-36), marital relationship (0-42). The child-related stress is described by adaptation (scores: 0-78), temperament (0-60), distractability (0-72), demandingness (0-60), positive reinforcement (0-48), acceptance (0-72). An algorithm converts the subscores and the total score to a descriptive classification of parental stress level (very low, low, below average, average, above average, high, very high). Special norms hold for clinical samples.
  Higher values correspond to higher parental stress. A score reduction is a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Roeyers, Prof. dr., Principal Investigator — UGent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No